CLINICAL TRIAL: NCT05463744
Title: A Phase 3, Multicenter, Randomized, Parallel-Design, Open-Label Study to Evaluate the Efficacy and Safety of LY3209590 as a Weekly Basal Insulin Compared With Insulin Degludec in Participants With Type 1 Diabetes Treated With Multiple Daily Injection Therapy
Brief Title: A Study of Insulin Efsitora Alfa (LY3209590) Compared With Insulin Degludec in Participants With Type 1 Diabetes Treated With Multiple Daily Injection Therapy
Acronym: QWINT-5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18263; I8H-MC-BDCY (Other: Eli Lilly and Company); 2021-005892-38 (EudraCT Number)
Record Dates: First submitted 2022-07-15; First posted 2022-07-19 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Type 1 Diabetes; Diabetes
Keywords: Type 1 Diabetes (T1D)
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Insulin Efsitora Alfa (Experimental): Participants who were treated with prestudy basal insulin and prandial insulin therapy (100 units per milliliter (U/mL) Insulin Lispro) received 500 U/mL of insulin efsitora alfa administered once weekly (QW) for 52 weeks as subcutaneous injection, followed by a 5-week safety follow-up.
  Interventions: Drug: Insulin Efsitora Alfa
- Insulin Degludec (Active Comparator): Participants who were treated with prestudy basal insulin and prandial insulin therapy (100 U/mL Insulin Lispro) received 100 U/mL of Insulin Degludec administered once daily (QD) for 52 weeks as subcutaneous injection, followed by a 5-week safety follow-up.
  Interventions: Drug: Insulin Degludec

INTERVENTIONS:
Drug: Insulin Efsitora Alfa — Administered SC
  Other Names: LY3209590 and Basal Insulin-FC
  Arms: Insulin Efsitora Alfa
Drug: Insulin Degludec — Administered SC
  Arms: Insulin Degludec

SUMMARY:
The main purpose of this study is to measure the safety and efficacy of insulin efsitora alfa (LY3209590) compared with insulin degludec in participants with type 1 diabetes treated with multiple daily injection therapy.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of type 1 diabetes for at least 1 year prior to screening
* Have received treatment with basal-bolus insulin analog multiple daily injection therapy according to the local product label for at least 90 days prior to screening
* Have an HbA1c value of 7.0% to 10.0%, inclusive, as determined by the central laboratory at screening.
* Have a body mass index of ≤35 kilogram/square meter (kg/m²)

Exclusion Criteria:

* Have a diagnosis of type 2 diabetes, latent autoimmune diabetes, or specific types of diabetes other than type 1 diabetes
* Have a history of more than 1 episode of severe hypoglycemia, within the 6 months prior to screening.
* Have a history of more than 1 episode of diabetic ketoacidosis or hyperosmolar state or coma requiring hospitalization within the 6 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 692 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST, Study Chair — Eli Lilly and Company
Locations (83):
- United States (34):
  - John Muir Physician Network Research Center, Concord, California
  - Valley Research, Fresno, California
  - Catalina Research Institute, LLC, Montclair, California
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - University Clinical Investigators, Inc., Tustin, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Northeast Research Institute (NERI), Fleming Island, Florida
  - Jellinger and Lerman, MD PA dba The Center for Diabetes and Endocrine Care, Fort Lauderdale, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Hanson Clinical Research Center, Port Charlotte, Florida
  - East Coast Institute for Research at The Jones Center, Macon, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - MedStar Health Research Institute (MedStar Physician Based Research Network), Hyattsville, Maryland
  - Endocrine and Metabolic Consultants, Rockville, Maryland
  - Clinvest Research LLC, Springfield, Missouri
  - Palm Research Center Tenaya, Las Vegas, Nevada
  - Palm Research Center Sunset, Las Vegas, Nevada
  - Research Foundation of SUNY - University of Buffalo, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - NYC Research, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - Dallas Diabetes Research Center, Dallas, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - Research Institute of Dallas, Dallas, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Amir A Hassan, MD, PA, Houston, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - Texas Diabetes & Endocrinology, P.A., Round Rock, Texas
  - Rainier Clinical Research Center, Renton, Washington
- Argentina (14):
  - CEDIC, CABA, Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Ciudad Autónoma de Buenos Aire, Buenos Aires
  - Consultorio de Investigación Clínica EMO SRL, Ciudad Autonoma de Buenos Aire, Buenos Air
  - CIAD Moron, Morón, Buenos Air
  - Investigaciones Medicas Imoba Srl, Balvanera, Ciudad Autónoma de Buenos Aire
  - Mautalen Salud e Investigación, Buenos Aires, Ciudad Autónoma de Buenos Aire
  - Centro Medico Privado CEMAIC, Capital, Córdoba Province
  - Centro Medico Privado San Vicente Diabetes, Córdoba, Córdoba Province
  - Centro de Salud e Investigaciones Médicas, Santa Rosa, La Pampa Province
  - CIPADI - Centro Integral de Prevencion y Atencion en Diabetes, Godoy Cruz, Mendoza Province
  - Clínica Mayo de Urgencias Médicas Cruz Blanca S.R.L, San Miguel de Tucumán, Tucumán Province
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán, Tucumán Province
  - Instituto Médico Especializado (IME), Buenos Aires
  - Centro Diabetológico Dr. Waitman, Córdoba
- Japan (14):
  - Tosaki Clinic for Diabetes and Endocrinology, Nagoya, Aichi-ken
  - Manda Memorial Hospital, Sapporo, Hokkaido
  - MinamiAkatsukaClinic, Mito, Ibaraki
  - Nakakinen clinic, Naka, Ibaraki
  - Noritake Clinic, Ushiku, Ibaraki
  - Takai Internal Medicine Clinic, Kamakura-shi, Kanagawa
  - Takatsuki Red Cross Hospital, Takatsuki, Osaka
  - Shimizu Clinic Fusa, Saitama-shi, Saitama
  - The Institute for Adult Disease, Asahi Life Foundation, Chuo-ku, Tokyo
  - Hachioji Diabetes Clinic, Hachioji-shi, Tokyo
  - Clinic Masae Minami, Fukuoka
  - Jinnouchi Hospital, Kumamoto
  - Heiwadai Hospital, Miyazaki
  - Abe Clinic, Ōita
- Poland (10):
  - Medyczne Centrum Diabetologiczno Endokrynologiczno Metaboliczne DIAB-ENDO-MET, Krakow, Lesser Poland Voivodeship
  - Gabinety TERPA, Lublin, Lublin Voivodeship
  - NZOZ Medica, Lublin, Lublin Voivodeship
  - Centrum Medyczne "Diabetika", Radom, Masovian Voivodeship
  - Centralny Szpital Kliniczny MSWiA w Warszawie, Warsaw, Masovian Voivodeship
  - NBR Polska, Warsaw, Mazowiecki
  - SN ZOZ Lege Artis Poradnia Diabetologiczna, Bialystok, Podlaskie Voivodeship
  - NZOZ Specjalistyczny Ośrodek Internistyczno-Diabetologiczny, Bialystok, Podlaskie Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
  - Private Practice - Dr. Janusz Gumprecht, Zabrze, Silesian Voivodeship
- Puerto Rico (2):
  - Advanced Clinical Research, LLC, Bayamón
  - Endocrinologist Metabolic Clinic & Research Institute, San Juan
- Slovakia (3):
  - Tatratrial s.r.o., Rožňava, Košice Region
  - Funkystuff, Nové Zámky, Nitra Region
  - ENDIAMED s.r.o, Dolný Kubín, Žilina Region
- Taiwan (6):
  - Chung Shan Medical University Hospital, Taichung, Taichung
  - Taichung Veterans General Hospital, Taichung, Taichung
  - Chi Mei Medical Center, Tainan, Tainan
  - Taipei Veterans General Hospital, Taipei City, Taipei
  - Changhua Christian Hospital, Changhua
  - National Cheng Kung University Hospital, Tainan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Bergenstal RM, Weinstock RS, Mathieu C, Onishi Y, Vijayanagaram V, Katz ML, Carr MC, Chang AM. Once-weekly insulin efsitora alfa versus once-daily insulin degludec in adults with type 1 diabetes (QWINT-5): a phase 3 randomised non-inferiority trial. Lancet. 2024 Sep 21;404(10458):1132-1142. doi: 10.1016/S0140-6736(24)01804-X. Epub 2024 Sep 10. PMID 39270686
- See also: A Study of LY3209590 Compared With Insulin Degludec in Participants With Type 1 Diabetes Treated With Multiple Daily Injection Therapy (QWINT-5) — https://trials.lilly.com/en-US/trial/351115

RESULTS

PARTICIPANT FLOW:
Groups:
- 500 U/mL Insulin Efsitora Alfa: Participants who were treated with prestudy basal insulin and prandial insulin therapy (100 units per milliliter (U/mL) Insulin Lispro) received 500 U/mL of insulin efsitora alfa administered once weekly (QW) for 52 weeks as subcutaneous injection, followed by a 5-week safety follow-up.
- 100 U/mL Insulin Degludec: Participants who were treated with prestudy basal insulin and prandial insulin therapy (100 U/mL Insulin Lispro) received 100 U/mL of Insulin Degludec administered once daily (QD) for 52 weeks as subcutaneous injection, followed by a 5-week safety follow-up.
Period: Treatment Period
Arm/Group | 500 U/mL Insulin Efsitora Alfa | 100 U/mL Insulin Degludec
Started | 343 | 349
Received at Least One Dose of Study Drug | 343 | 349
Completed | 316 | 319
Not Completed | 27 | 30
Not completed — Withdrawal by Subject | 19 | 16
Not completed — Adverse Event | 4 | 4
Not completed — Pregnancy | 0 | 3
Not completed — Lost to Follow-up | 1 | 3
Not completed — Inadvertent enrollment | 2 | 1
Not completed — Death | 0 | 1
Not completed — Non-compliance with Study Drug | 1 | 0
Not completed — Subject Terminated by Sponsor | 0 | 1
Not completed — Physician Decision | 0 | 1
Period: Follow-Up Period
Arm/Group | 500 U/mL Insulin Efsitora Alfa | 100 U/mL Insulin Degludec
Started | 332 (Per statistical analysis plan, participants who completed the study treatment period were required to complete a safety follow-up period and participants who discontinued the study treatment prematurely were encouraged to remain in the study for safety monitoring.) | 326 (Per statistical analysis plan, participants who completed the study treatment period were required to complete a safety follow-up period and participants who discontinued the study treatment prematurely were encouraged to remain in the study for safety monitoring.)
Completed | 328 | 324
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of the study drug.
Groups:
- 500 U/mL Insulin Efsitora Alfa: Participants who were treated with prestudy basal insulin and prandial insulin therapy (100 U/mL) Insulin Lispro) received 500 U/mL of insulin efsitora alfa administered once weekly (QW) for 52 weeks as subcutaneous injection, followed by a 5-week safety follow-up
- 100 U/mL Insulin Degludec: Participants who were treated with prestudy basal insulin and prandial insulin therapy (100 U/mL Insulin Lispro) received 100 U/mL of Insulin Degludec administered QD for 52 weeks as subcutaneous injection, followed by a 5-week safety follow-up.
- Total: Total of all reporting groups
Arm/Group | 500 U/mL Insulin Efsitora Alfa | 100 U/mL Insulin Degludec | Total
Number analyzed (Participants) | 343 | 349 | 692
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.40 (14.22) | 43.60 (14.01) | 44.00 (14.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 158 | 308
  Male | 193 | 191 | 384
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 121 | 116 | 237
  Not Hispanic or Latino | 221 | 230 | 451
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 69 | 73 | 142
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 11 | 13 | 24
  White | 259 | 262 | 521
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 98 | 99 | 197
  Japan | 48 | 53 | 101
  Poland | 66 | 66 | 132
  Slovakia | 15 | 17 | 32
  Taiwan | 15 | 17 | 32
  United States | 101 | 97 | 198
HemoglobinA1c (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycosylated fraction of hemoglobin A. It is measured primarily to identify the average plasma glucose concentration over prolonged periods of time.
  Percentage of HbA1c | 7.88 (0.75) | 7.94 (0.72) | 7.91 (0.73)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at Week 26 [Noninferiority Analysis]
Description: HbA1c is the glycosylated fraction of hemoglobin A. It is measured primarily to identify the average plasma glucose concentration over prolonged periods of time.
  Least Squares (LS) mean was determined using Analysis of Covariance (ANCOVA) model with treatment + country + CGM use prior to study entry [yes/no]+ carbohydrate counting for prandial insulin[yes/no] + baseline value of the dependent variable (Type III sum of squares) as variables. Missing data at Week 26 were imputed by return-to-baseline multiple imputations approach.
Time Frame: Baseline, Week 26
Population: All randomized participants who received at least one dose of the study drug and had HbA1c measurement at baseline or Week 26. Participants who discontinued the study drug due to inadvertent enrollment were excluded.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Groups:
- 500 U/mL Insulin Efsitora Alfa: Participants who are treated with prestudy basal insulin and prandial insulin therapy (100 U/mL) Insulin Lispro) received 500 U/mL of insulin efsitora alfa administered once weekly (QW) for 52 weeks as subcutaneous injection, followed by a 5-week safety follow-up
- 100 U/mL Insulin Degludec: Participants who are treated with prestudy basal insulin and prandial insulin therapy (100 U/mL Insulin Lispro) received 100 U/mL of Insulin Degludec administered QD for 52 weeks as subcutaneous injection, followed by a 5-week safety follow-up.
Arm/Group | 500 U/mL Insulin Efsitora Alfa | 100 U/mL Insulin Degludec
Number analyzed (Participants) | 341 | 348
Percentage of HbA1c | -0.51 (0.0469) | -0.56 (0.0463)
Statistical Analysis 1: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Test type: Non-Inferiority — 0.4% noninferiority margin (NIM); ANCOVA; LS Mean Difference = 0.052, 95% CI 2-sided [-0.077 to 0.181]

2. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at Week 26 [Superiority Analysis]
Description: HbA1c is the glycosylated fraction of hemoglobin A. It is measured primarily to identify the average plasma glucose concentration over prolonged periods of time.
  LS mean was determined using ANCOVA model with treatment + country + CGM use prior to study entry [yes/no] + carbohydrate counting for prandial insulin[yes/no] + baseline value of the dependent variable (Type III sum of squares) as variables. Missing data at Week 26 were imputed by return-to-baseline multiple imputations approach.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 500 U/mL Insulin Efsitora Alfa | 100 U/mL Insulin Degludec
Number analyzed (Participants) | 341 | 348
Percentage of HbA1c | -0.51 (0.0469) | -0.56 (0.0463)
Statistical Analysis 1: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Test type: Superiority; p = 0.432, ANCOVA; LS Mean Difference = 0.052, 95% CI 2-sided [-0.077 to 0.181]

3. Secondary Outcome: Percentage of Time in the Blood Glucose Range Between 70 and 180 mg/dL [3.9 and 10.0 mmol/L] From Week 23 to Week 26
Description: Percentage of time in glucose range between 70 and 180 milligram per deciliter (mg/dL) [3.9 and 10.0 millimole per liter (mmol/L)], measured by continued glucose monitoring (CGM) from week 23 to week 26 inclusive over a 24-Hour Period. The time component of the time-in-range statistic was calculated using the display time recorded by the CGM device.
  LS mean was determined using ANCOVA model with treatment + country + CGM use prior to study entry [yes/no] + carbohydrate counting for prandial insulin dosing [yes/no] + Hemoglobin A1c Stratum at Baseline and baseline value of the dependent variable (Type III sum of squares) as variables. Missing data at Week 23-26 were imputed by return-to-baseline multiple imputations approach
Time Frame: Week 23 to Week 26
Population: All randomized participants who took at least one dose of the study drug and had evaluable data for this outcome at baseline or Week 23-26 were included. Participants who discontinued the study drug due to inadvertent enrollment were excluded.
Measure: Least Squares Mean (Standard Error); unit: Percentage of time
Groups:
- 500 U/mL Insulin Efsitora Alfa: Participants who are treated with prestudy basal insulin and prandial insulin therapy (100 U/mL Insulin Lispro) received 500 U/mL of insulin efsitora alfa administered QW for 52 weeks as subcutaneous injection, followed by a 5-week safety follow-up.
Arm/Group | 500 U/mL Insulin Efsitora Alfa | 100 U/mL Insulin Degludec
Number analyzed (Participants) | 339 | 347
Percentage of time | 52.54 (0.691) | 52.85 (0.684)
Statistical Analysis 1: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Test type: Superiority; p = 0.751, ANCOVA; LS Mean Difference = -0.31, 95% CI 2-sided [-2.22 to 1.60]

4. Secondary Outcome: Nocturnal Hypoglycemia Event Rate
Description: The event rate of participant-reported clinically significant nocturnal hypoglycemia (defined as blood glucose level <54 mg/dL (3.0 mmol/L) or severe hypoglycemia and occurs at night and presumably during sleep between midnight and 6:00 AM), measured during treatment phase up to week 52.
  Group mean was reported and determined by Negative binomial model using Number of episodes = Baseline hypoglycemia rate + HbA1c at Baseline (%) + Treatment, with log (exposure in days/365.25) as an offset variable.
Time Frame: Baseline up to Week 52
Population: All randomized participants who received at least one dose of the study drug and had evaluable data for this outcome.
Measure: Mean (Standard Error); unit: events per year
Arm/Group | 500 U/mL Insulin Efsitora Alfa | 100 U/mL Insulin Degludec
Number analyzed (Participants) | 343 | 349
events per year | 1.99 (0.180) | 1.96 (0.177)
Statistical Analysis 1: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Test type: Superiority; p = 0.900, Negative binomial model; Relative Rate = 1.02, 95% CI 2-sided [0.79 to 1.31]

5. Secondary Outcome: Change From Baseline in HbA1c at Week 52 [Noninferiority Analysis]
Description: HbA1c is the glycosylated fraction of hemoglobin A. It is measured primarily to identify the average plasma glucose concentration over prolonged periods of time.
  LS mean was determined using ANCOVA model with treatment + country + CGM use prior to study entry [yes/no]+ carbohydrate counting for prandial insulin[yes/no] + baseline value of the dependent variable (Type III sum of squares) as variables. Missing data at Week 52 were imputed by return-to-baseline multiple imputations approach
Time Frame: Baseline, Week 52
Population: All randomized participants who received at least one dose of the study drug and had HbA1c measurement at baseline or Week 52. Participants who discontinued the study drug due to inadvertent enrollment were excluded.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | 500 U/mL Insulin Efsitora Alfa | 100 U/mL Insulin Degludec
Number analyzed (Participants) | 341 | 348
percentage of HbA1c | -0.38 (0.0484) | -0.40 (0.0479)
Statistical Analysis 1: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Test type: Non-Inferiority — 0.4% noninferiority margin (NIM); ANCOVA; LS Mean Difference = 0.024, 95% CI 2-sided [-0.110 to 0.157], Standard Error of Mean 0.0682

6. Secondary Outcome: Change From Baseline in Fasting Blood Glucose
Description: Change from baseline in fasting blood glucose measured by self-monitoring blood glucose (SMBG).
  LS mean was determined using ANCOVA model with treatment, country, CGM use prior to study entry [yes/no], carbohydrate counting for prandial insulin dosing [yes/no]) and baseline value of the dependent variable as variables. Missing data at Baseline were imputed with multiple imputation with assumption of missing at random. Missing data were imputed by return-to-baseline multiple imputations approach.
Time Frame: Baseline, Week 26, and Week 52
Population: All randomized participants who received at least one dose of the study drug and had evaluable data for this outcome at Baseline, Week 26, or Week 52 were included in the analysis. For the Week 26 analysis, data from Baseline or Week 26 were considered, while for the Week 52 analysis, data from Baseline or Week 52 were included. Participants who discontinued the study drug due to inadvertent enrollment were excluded.
Measure: Least Squares Mean (Standard Error); unit: milligram per deciliter (mg/dL)
Arm/Group | 500 U/mL Insulin Efsitora Alfa | 100 U/mL Insulin Degludec
Number analyzed (Participants) | 341 | 348
milligram per deciliter (mg/dL)
  Week 26 | -26.67 (2.247) | -25.45 (2.222)
  Week 52 | -24.78 (2.478) | -19.93 (2.452)
Statistical Analysis 1: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Week 26; Test type: Superiority; p = 0.697, ANCOVA; LS Mean Difference = -1.22, 95% CI 2-sided [-7.38 to 4.93]
Statistical Analysis 2: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Week 52; Test type: Superiority; p = 0.163, ANCOVA; LS Mean Difference = -4.84, 95% CI 2-sided [-11.64 to 1.96]

7. Secondary Outcome: Glucose Variability
Description: Glucose variability measured as coefficient of variation (CV) for blood glucose during the CGM session over a 24-hour period, between Week 23 to Week 26 and Week 49 to Week 52 was reported.
  LS mean was determined using mixed model repeated measures (MMRM) model with BASELINE + Country + Prior CGM use + Carbohydrate counting for Prandial Dose + Hemoglobin A1c Stratum at Baseline + Treatment + Time + Treatment*Time (Type III sum of squares) as variables. Unstructured variance-covariance structure was used.
Time Frame: Week 23 to Week 26 and Week 49 to Week 52
Population: All randomized participants who took at least one dose of the study drug and had a baseline and at least one post- baseline value for this outcome. Participants who discontinued the study drug due to inadvertent enrollment were excluded
Measure: Least Squares Mean (Standard Error); unit: percentage of CV
Arm/Group | 500 U/mL Insulin Efsitora Alfa | 100 U/mL Insulin Degludec
Number analyzed (Participants) | 331 | 332
percentage of CV
  Week 23 to Week 26 | 33.72 (0.230) | 33.69 (0.229)
  Week 49 to Week 52 | 33.69 (0.233) | 33.18 (0.233)
Statistical Analysis 1: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Week 23 to Week 26; Test type: Superiority; p = 0.939, Mixed Models Analysis; LS Mean Difference = 0.02, 95% CI 2-sided [-0.61 to 0.66]
Statistical Analysis 2: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Week 49 to Week 52; Test type: Superiority; p = 0.116, Mixed Models Analysis; LS Mean Difference = 0.52, 95% CI 2-sided [-0.13 to 1.17]

8. Secondary Outcome: Percentage of Time in the Blood Glucose Range Between 70 and 180 mg/dL [3.9 and 10.0 mmol/L] From Week 49 to Week 52
Description: Percentage of time spent within the blood glucose range of 70 to 180 mg/dL [3.9 to 10.0 mmol/L], as measured during the CGM session over a 24-hour period, from Week 49 to Week 52.
  LS mean was determined using ANCOVA model with treatment, country, CGM use prior to study entry [yes/no], carbohydrate counting for prandial insulin dosing [yes/no]) and Hemoglobin A1c Stratum at baseline and baseline value of the dependent variable as variables. Missing data at Baseline were imputed with multiple imputation with assumption of missing at random. Missing data were imputed by return-to-baseline multiple imputations approach.
Time Frame: Week 49 to Week 52
Population: All randomized participants who received at least one dose of the study drug and had evaluable data for this outcome at baseline or Week 49-52 were included in the analysis. Participants who discontinued the study drug due to inadvertent enrollment were excluded.
Measure: Least Squares Mean (Standard Error); unit: percentage of time
Arm/Group | 500 U/mL Insulin Efsitora Alfa | 100 U/mL Insulin Degludec
Number analyzed (Participants) | 338 | 347
percentage of time | 50.28 (0.755) | 49.74 (0.744)
Statistical Analysis 1: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Test type: Superiority; p = 0.610, ANCOVA; LS Mean Difference = 0.54, 95% CI 2-sided [-1.54 to 2.62]

9. Secondary Outcome: Basal Insulin Dose
Description: The insulin dose was recorded daily or weekly in an electronic diary. The average weekly basal insulin dose at Week 26 and Week 52 was reported.
  LS mean was determined using MMRM model with BASELINE + Hemoglobin A1c Stratum at Baseline + Country + Prior CGM use + Carbohydrate counting for Prandial Dose + Treatment + Time + Treatment*Time (Type III sum of squares) as variables. Variance-covariance structure was set as compound symmetry.
Time Frame: Week 26 and Week 52
Population: All randomized participants who received at least one dose of the study drug and had a baseline and at least one post-baseline value for this outcome. Participants who discontinued the study drug due to inadvertent enrollment were excluded.
Measure: Least Squares Mean (Standard Error); unit: Units per week (U/week)
Arm/Group | 500 U/mL Insulin Efsitora Alfa | 100 U/mL Insulin Degludec
Number analyzed (Participants) | 341 | 347
Units per week (U/week)
  Week 26 | 199.51 (4.47) | 208.47 (4.43)
  Week 52 | 204.37 (4.50) | 211.25 (4.46)
Statistical Analysis 1: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Week 26; Test type: Superiority; p = 0.155, Mixed Models Analysis; LS Mean Difference = -8.96, 95% CI 2-sided [-21.30 to 3.38]
Statistical Analysis 2: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Week 52; Test type: Superiority; p = 0.278, Mixed Models Analysis; LS Mean Difference = -6.88, 95% CI 2-sided [-19.31 to 5.55]

10. Secondary Outcome: Bolus Insulin Dose
Description: The insulin dose was recorded daily or weekly in an electronic diary. The average daily bolus insulin dose at Week 26 and Week 52 was reported.
  LS mean was determined using MMRM model with BASELINE + Hemoglobin A1c Stratum at Baseline + Country + Prior CGM use + Carbohydrate counting for Prandial Dose + Treatment + Time + Treatment*Time (Type III sum of squares) as variables. Variance-covariance structure was set as compound symmetry.
Time Frame: Week 26 and Week 52
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Units per day (U/day)
Arm/Group | 500 U/mL Insulin Efsitora Alfa | 100 U/mL Insulin Degludec
Number analyzed (Participants) | 307 | 327
Units per day (U/day)
  Week 26 | 21.48 (0.64) | 25.25 (0.62)
  Week 52 | 22.62 (0.65) | 26.10 (0.63)
Statistical Analysis 1: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Week 26; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -3.77, 95% CI 2-sided [-5.52 to -2.03]
Statistical Analysis 2: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Week 52; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -3.49, 95% CI 2-sided [-5.26 to -1.71]

11. Secondary Outcome: Total Insulin Dose
Description: The average weekly total insulin dose is the sum of the average weekly basal and bolus doses. LS mean was determined using MMRM model with BASELINE + Hemoglobin A1c Stratum at Baseline + Country + Prior CGM use + Carbohydrate counting for Prandial Dose + Treatment + Time + Treatment*Time (Type III sum of squares) as variables. Variance-covariance structure was set as compound symmetry.
Time Frame: Week 26 and Week 52
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Units per week (U/week)
Arm/Group | 500 U/mL Insulin Efsitora Alfa | 100 U/mL Insulin Degludec
Number analyzed (Participants) | 305 | 327
Units per week (U/week)
  Week 26 | 343.91 (6.72) | 383.19 (6.47)
  Week 52 | 355.66 (6.81) | 391.60 (6.53)
Statistical Analysis 1: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Week 26; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -39.28, 95% CI 2-sided [-57.59 to -20.98]
Statistical Analysis 2: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Week 52; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -35.94, 95% CI 2-sided [-54.44 to -17.43]

12. Secondary Outcome: Basal Insulin Dose to Total Insulin Dose Ratio
Description: The basal/total insulin dose ratio is the average weekly basal dose divided by the average weekly total dose.
  LS mean was determined using MMRM model with BASELINE + Hemoglobin A1c Stratum at Baseline + Country + Prior CGM use + Carbohydrate counting for Prandial Dose + Treatment + Time + Treatment*Time (Type III sum of squares) as variables. Variance-covariance structure was set as compound symmetry.
Time Frame: Week 26 and Week 52
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Percentage of basal/total insulin dose
Arm/Group | 500 U/mL Insulin Efsitora Alfa | 100 U/mL Insulin Degludec
Number analyzed (Participants) | 305 | 327
Percentage of basal/total insulin dose
  Week 26 | 56.4 (0.69) | 53.2 (0.66)
  Week 52 | 55.4 (0.70) | 52.6 (0.67)
Statistical Analysis 1: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Week 26; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = 3.19, 95% CI 2-sided [1.32 to 5.06]
Statistical Analysis 2: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Week 52; Test type: Superiority; p = 0.004, Mixed Models Analysis; LS Mean Difference = 2.80, 95% CI 2-sided [0.91 to 4.70]

13. Secondary Outcome: Hypoglycemia Event Rate
Description: Rate of Composite Level 2 and 3 Hypoglycemia Events were reported. Hypoglycemia with glucose <54 mg/dL (Level 2) or Severe Hypoglycemia confirmed by the investigator to be an event that required assistance for treatment (Level 3) was reported. A severe hypoglycemic event is characterized by altered mental or physical status requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions for the treatment of hypoglycemia.
  Group mean was reported and determined by Negative binomial model using Number of episodes = Baseline hypoglycemia rate + HbA1c at Baseline (%) + Treatment, with log (exposure in days/365.25) as an offset variable.
Time Frame: Baseline up to Week 52
Population: All randomized participants who received at least one dose of the study drug.
Measure: Mean (Standard Error); unit: Events per year
Arm/Group | 500 U/mL Insulin Efsitora Alfa | 100 U/mL Insulin Degludec
Number analyzed (Participants) | 343 | 349
Events per year | 14.03 (0.816) | 11.59 (0.681)
Statistical Analysis 1: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Test type: Superiority; p = 0.016, Negative binomial model; Relative Rate = 1.21, 95% CI 2-sided [1.04 to 1.41]

14. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight was reported. LS Mean was determined by MMRM model using Baseline + Treatment + Time + Treatment*Time (Type III sum of squares) as variables. Variance-covariance structure was set as compound symmetry.
Time Frame: Baseline, Week 26, and Week 52
Population: All randomized participants who received at least one dose of the study drug and had baseline, at least one post-baseline evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | 500 U/mL Insulin Efsitora Alfa | 100 U/mL Insulin Degludec
Number analyzed (Participants) | 342 | 348
kilograms (kg)
  Week 26 | 1.71 (0.159) | 1.62 (0.158)
  Week 52 | 1.96 (0.160) | 1.85 (0.159)
Statistical Analysis 1: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Week 26; Test type: Superiority; p = 0.702, Mixed Models Analysis; LS Mean Difference = 0.086, 95% CI 2-sided [-0.35 to 0.53]
Statistical Analysis 2: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Week 52; Test type: Superiority; p = 0.609, Mixed Models Analysis; LS Mean Difference = 0.12, 95% CI 2-sided [-0.33 to 0.56]

15. Secondary Outcome: Percentage of Time in Hypoglycemia Range With Blood Glucose <54 mg/dL (3.0 mmol/L)
Description: Percentage of time spent in the hypoglycemia range with blood glucose < 54 mg/dL (3.0 mmol/L), as measured during the CGM session over a 24-hour period from week 23 to week 26 and week 49 to week 52 was reported. LS Mean was determined by ANCOVA model using treatment + country + CGM use prior to study entry [yes/no] + carbohydrate counting for prandial insulin dosing [yes/no] + Hemoglobin A1c Stratum at Baseline and baseline value of the dependent variable (Type III sum of squares). as variables. Missing data at Baseline were imputed with multiple imputation with assumption of missing at random. Missing data at week 23-26 and week 49-52 were imputed by return-to-baseline multiple imputations approach.
Time Frame: Week 23 to Week 26 and Week 49 to Week 52
Population: All randomized participants who received at least one dose of the study drug and had evaluable data for this outcome at Baseline, Week 23-26, or Week 49-52 were included in the analysis. For the Week 23-26 analysis, data from Baseline or Week 23-26 were considered, while for the Week 49-52 analysis, data from Baseline or Week 49-52 were included. Participants who discontinued the study drug due to inadvertent enrollment were excluded.
Measure: Least Squares Mean (Standard Error); unit: percentage of time
Arm/Group | 500 U/mL Insulin Efsitora Alfa | 100 U/mL Insulin Degludec
Number analyzed (Participants) | 339 | 347
percentage of time
  Week 23 to Week 26 | 0.75 (0.058) | 0.72 (0.057)
  Week 49 to Week 52 | 0.74 (0.053) | 0.64 (0.052)
Statistical Analysis 1: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Week 23 to Week 26; Test type: Superiority; p = 0.681, ANCOVA; LS Mean Difference = 0.03, 95% CI 2-sided [-0.13 to 0.19]
Statistical Analysis 2: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Week 49 to Week 52; Test type: Superiority; p = 0.182, ANCOVA; LS Mean Difference = 0.10, 95% CI 2-sided [-0.05 to 0.24]

16. Secondary Outcome: Percentage of Time in Hyperglycemia Range With Blood Glucose >180 mg/dL (10.0 mmol/L) From Week 23 to Week 26
Description: Percentage of time spent in the hyperglycemia range with blood glucose greater than (>) 180 mg/dL (10.0 mmol/L), as measured during the CGM session over a 24-hour period from Week 23 to Week 26 was reported.
  LS Mean was determined by ANCOVA model using treatment + country + CGM use prior to study entry [yes/no] + carbohydrate counting for prandial insulin dosing [yes/no] + Hemoglobin A1c Stratum at Baseline and baseline value of the dependent variable (Type III sum of squares) as variables. Missing data at Baseline were imputed with multiple imputation with assumption of missing at random. Missing data at week 23-week 26 were imputed by return-to-baseline multiple imputations approach.
Time Frame: Week 23 to Week 26
Population: All randomized participants who received at least one dose of the study drug and had evaluable data for this outcome at baseline or Week 23-26 were included in the analysis. Participants who discontinued the study drug due to inadvertent enrollment were excluded
Measure: Least Squares Mean (Standard Error); unit: percentage of time
Arm/Group | 500 U/mL Insulin Efsitora Alfa | 100 U/mL Insulin Degludec
Number analyzed (Participants) | 339 | 347
percentage of time | 44.29 (0.743) | 44.29 (0.735)
Statistical Analysis 1: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Week 23 to Week 26; Test type: Superiority; p = 0.999, ANCOVA; LS Mean Difference = -0.00, 95% CI 2-sided [-2.06 to 2.05]

17. Secondary Outcome: Percentage of Time in Hyperglycemia Range With Blood Glucose >180 mg/dL (10.0 mmol/L) From Week 49 to Week 52
Description: Percentage of time spent in the hyperglycemia range with blood glucose greater than (>) 180 mg/dL (10.0 mmol/L), as measured during the CGM session over a 24-hour period from Week 49 to Week 52 was reported.
  LS Mean was determined by ANCOVA model using treatment + country + CGM use prior to study entry [yes/no] + carbohydrate counting for prandial insulin dosing [yes/no] + Hemoglobin A1c Stratum at Baseline and baseline value of the dependent variable (Type III sum of squares) as variables. Missing data at Baseline were imputed with multiple imputation with assumption of missing at random. Missing data at week 49-week 52 were imputed by return-to-baseline multiple imputations approach.
Time Frame: Week 49 to Week 52
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: percentage of time
Arm/Group | 500 U/mL Insulin Efsitora Alfa | 100 U/mL Insulin Degludec
Number analyzed (Participants) | 338 | 347
percentage of time | 46.73 (0.811) | 47.56 (0.797)
Statistical Analysis 1: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Test type: Superiority; p = 0.468, ANCOVA; LS Mean Difference = -0.83, 95% CI 2-sided [-3.06 to 1.41]

18. Secondary Outcome: Diabetes Treatment Satisfaction as Measured by the Diabetes Treatment Satisfaction Questionnaire, Change Version (DTSQc) at Week 26
Description: The Diabetes Treatment Satisfaction Questionnaire change (DTSQc) score is used to assess relative change in participant satisfaction from baseline. The questionnaire consists of 8 items, 6 of which measure Treatment Satisfaction, dealing with: 1. satisfaction with current treatment; 2. convenience of the treatment; 3. flexibility; 4. satisfaction with own understanding of participant's diabetes; 5. how likely to recommend their present treatment; and 6. how satisfied to continue with their present treatment. Each item is rated on a 7-point Likert scale (which ranges from -3 (much less satisfied) to +3 (much more satisfied). The scores from the 6 treatment satisfaction items are summed to a Total Treatment Satisfaction Score, which ranges from -18 (much less satisfied) to +18 (much more satisfied). Higher the score the greater the improvement in satisfaction with treatment. The lower the score the greater the deterioration in satisfaction with treatment.
Time Frame: Week 26
Population: All randomized participants who received at least one dose of the study drug and had evaluable data for this outcome. Participants who discontinued the study drug due to inadvertent enrollment were excluded.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 500 U/mL Insulin Efsitora Alfa | 100 U/mL Insulin Degludec
Number analyzed (Participants) | 306 | 314
score on a scale | 14.4 (4.53) | 13.2 (5.20)
Statistical Analysis 1: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Test type: Other; p = 0.008, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Diabetes Treatment Satisfaction as Measured by the Diabetes Treatment Satisfaction Questionnaire, Change Version (DTSQc) at Week 52
Description: The DTSQc score is used to assess relative change in participant satisfaction from baseline. The questionnaire consists of 8 items, 6 of which measure Treatment Satisfaction, dealing with: 1. satisfaction with current treatment; 2. convenience of the treatment; 3. flexibility; 4. satisfaction with own understanding of participant's diabetes; 5. how likely to recommend their present treatment; and 6. how satisfied to continue with their present treatment. Each item is rated on a 7-point Likert scale (which ranges from -3 (much less satisfied) to +3 (much more satisfied). The scores from the 6 treatment satisfaction items are summed to a Total Treatment Satisfaction Score, which ranges from -18 (much less satisfied) to +18 (much more satisfied). Higher the score the greater the improvement in satisfaction with treatment. The lower the score the greater the deterioration in satisfaction with treatment.
Time Frame: Week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 500 U/mL Insulin Efsitora Alfa | 100 U/mL Insulin Degludec
Number analyzed (Participants) | 310 | 312
score on a scale | 14.4 (5.31) | 12.8 (5.67)
Statistical Analysis 1: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Change From Baseline in Short Form-36 Version 2 (SF-36 v2) Acute Form (Physical-Component and Mental-Component) Scores
Description: The SF-36v2 is a participant-reported measure designed to assess health status using 36 items across 8 domains: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. The 8 health domains are aggregated into two summary scores known as the physical component summary (PCS) score and the mental component summary (MCS) score. Scoring of each domain and both summary scores are norm based and presented in the form of T-scores, with a mean of 50 and a standard deviation of 10. Higher scores indicate better levels of function and/or better health. Range cannot be specified in norm-based scores.
  LS Mean was determined by MMRM model with Baseline + Country + Carbohydrate counting for Prandial Dose + Prior CGM use + Hemoglobin A1c Stratum at Baseline + Treatment + Time + Treatment*Time (Type III sum of squares). as variables. Unstructured variance-covariance structure was used.
Time Frame: Baseline, Week 26, and Week 52
Population: All randomized participants who received at least one dose of the study drug, had a baseline and at least one post- baseline value for this outcome. Participants who discontinued the study drug due to inadvertent enrollment were excluded.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | 500 U/mL Insulin Efsitora Alfa | 100 U/mL Insulin Degludec
Number analyzed (Participants) | 327 | 330
T-score
  Physical Component Score: Week 26 | 0.19 (0.275) | -0.24 (0.272)
  Physical Component Score: Week 52 | 0.48 (0.262) | -0.25 (0.260)
  Mental Component Score: Week 26 | 0.58 (0.419) | 0.36 (0.415)
  Mental Component Score: Week 52 | 0.61 (0.419) | 0.16 (0.417)
Statistical Analysis 1: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Physical Component Score: Week 26; Test type: Superiority; p = 0.270, Mixed Models Analysis; LS Mean Difference = 0.43, 95% CI 2-sided [-0.33 to 1.19]
Statistical Analysis 2: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Physical Component Score: Week 52; Test type: Superiority; p = 0.050, Mixed Models Analysis; LS Mean Difference = 0.73, 95% CI 2-sided [0.000 to 1.45]
Statistical Analysis 3: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Mental Component Score: Week 26; Test type: Superiority; p = 0.710, Mixed Models Analysis; LS Mean Difference = 0.22, 95% CI 2-sided [-0.94 to 1.38]
Statistical Analysis 4: Comparison: 500 U/mL Insulin Efsitora Alfa vs 100 U/mL Insulin Degludec; Mental Component Score: Week 52; Test type: Superiority; p = 0.447, Mixed Models Analysis; LS Mean Difference = 0.45, 95% CI 2-sided [-0.71 to 1.61]

ADVERSE EVENTS:
Time Frame: Baseline to end of safety follow-up (up to 57 weeks)
Description: All randomized participants who received at least one dose of study drug. Gender specific events occurring only in male or female participants have had the number of participants at risk adjusted accordingly.
  Participants were analyzed based on the actual treatment they received.
Arm/Group | 500 U/mL Insulin Efsitora Alfa | 100 U/mL Insulin Degludec
All-Cause Mortality (participants affected / at risk) | 0/343 | 1/349
Serious Adverse Events (participants affected / at risk) | 45/343 | 24/349
Other Adverse Events (participants affected / at risk) | 117/343 | 119/349
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 500 U/mL Insulin Efsitora Alfa (N=343) | 100 U/mL Insulin Degludec (N=349)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (2)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2)
Chronic granulomatous disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Limb reduction defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 27 (33) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic seizure (Nervous system disorders) | 1 (1) | 1 (1)
Hypoglycaemic unconsciousness (Nervous system disorders) | 10 (11) | 4 (5)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2/150 (2) | 0/158 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 500 U/mL Insulin Efsitora Alfa (N=343) | 100 U/mL Insulin Degludec (N=349)
Covid-19 (Infections and infestations) | 16 (16) | 23 (24)
Influenza (Infections and infestations) | 27 (30) | 18 (22)
Nasopharyngitis (Infections and infestations) | 40 (45) | 42 (54)
Upper respiratory tract infection (Infections and infestations) | 24 (29) | 30 (35)
Urinary tract infection (Infections and infestations) | 21 (24) | 11 (16)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 19 (20) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/44/NCT05463744/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT05463744/SAP_001.pdf